CLINICAL TRIAL: NCT02895763
Title: Development of a New Scale of Quality of Life, Specific of Neuro Muscular Diseases and More Specifically of Steinert Disease, by the Rasch Model Methods.
Brief Title: Quality of Life in Neuromuscular Disease
Acronym: QoLNMD
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2015Ao005
Record Dates: First submitted 2016-08-18; First posted 2016-09-12 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Quality of Life; Muscular Dystrophies
Keywords: QUALITY OF LIFE; NEUROMUSCULAR DISEASES
MeSH Terms: conditions — Muscular Dystrophies; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Neuro Muscular disease patients: French Patients, young adults and adults, with a diagnosed neuromuscular disease, of any known form.
  Interventions: Other: Form administrations

INTERVENTIONS:
Other: Form administrations

SUMMARY:
A Quality work was conducted to enable the future construction of a Quality of Life Questionnaire Related to Health (HRQoL) in patients with slowly progressive neuromuscular disease (NMD) as myopathies and muscular dystrophies. The discussion group training is an effective method to perform a thorough investigation of aspects of HRQoL potentially altered by NMD. Patients were recruited in France by 4 reference centers MNMs. All verbal interactions between participants focus groups were recorded. A qualitative analysis of the transcript was performed. The transcript provided 2424 CIF categories. The results helped to identify and quantify aspects of life that are altered by NMDs between patients. A pool of 64 items and a validated questionnaire (the WHOQOLBREF) were thern passed by 159 patients enrolled in eight reference centers MNMs. The investigators constructed a questionnaire called QoLNMD which is composed of two general items and 24 items classified into three areas: (1) \ Impact bodily symptoms, "(2) \ Self-perception" and (3) \ Activity participation. "Each area has good psychometric properties (Cronbach's alpha> 0.77, test-retest ICC> 0.81, H Loevinger> 0.41) and met the assumptions of IRT. the comparison with the WHOQOL-BREF was used to assess similarities and differences with a generic questionnaire. The next step was to validate the QoLNMD reassessing its psychometric properties in a new patient sample and calibrate the IRT measurement system. The purpose of these new part of study was to validate the French version of the QoL-NMD on a confirmatory sample of patients and to calibrate its measurement system. A prospective study in 8 NMD referral centers (France) was conducted. Both the QoL-NMD and a validated generic questionnaire (the WHOQOLBREF) were administered to patients. 156 patients were included for the confirmatory psychometric analysis. All three domains showed adequate psychometric properties and met IRT assumptions. The IRT model calibration was then performed successfully on 315 patients. The French version of the QoL-NMD showed adequate psychometric properties and can be used in rehabilitation services. A conversion table enables easy transformation of sum scores into IRT-calibrated measures. Minimum detectable change tables help interpreting score change.

DETAILED DESCRIPTION:
Quality work was conducted to enable the future construction of a Quality of Life Questionnaire Related to Health (HRQoL) in patients with slowly progressive neuromuscular disease (NMD) as myopathies and muscular dystrophies.

The discussion group training is an effective method to perform a thorough investigation of aspects of HRQoL potentially altered by NMD. Patients were recruited in France by 4 reference centers NMDs. To ensure that the performance in terms of severity would be adequate, three focus groups were formed: (1) Patients capable of walking. (2) Patients in wheelchairs. (3) Patients in wheelchairs and requiring continue ventilatory support. All verbal interactions between participants focus groups were recorded. A qualitative analysis of the transcript was performed according to the framework of the International Classification of Functioning, Disability and Health (ICF).

A total of 41 patients divided into five discussion groups were interviewed. The transcript provided 2424 ICF categories. References to percentages of different categories ICF were calculated and graphed.

The results helped to identify and quantify aspects of life that are altered by MNMs between patients. This qualitative work was the first phase of the ambitious project to develop a new specific questionnaire for NMDs HRQoL.

Build a questionnaire for assessing the quality of health-related life (HRQoL) in patients with NMD using item response theory (IRT).

A pool of 64 items and a validated questionnaire (the WHOQOLBREF) were passed by 159 patients enrolled in eight reference centers MNMs. The exploratory analysis included statistical methods derived from both the TRI and classical test theory.

The investigators constructed a questionnaire called QoLNMD which is composed of two general items and 24 items classified into three areas: (1) \ Impact bodily symptoms, "(2) \ Self-perception" and (3) \ Activity participation. "Each area has good psychometric properties (Cronbach's alpha> 0.77, test-retest ICC> 0.81, H Loevinger> 0.41) and met the assumptions of IRT. the comparison with the WHOQOL-BREF was used to assess similarities and differences with a generic questionnaire.

This study has allowed the development of a new HRQL questionnaire specifically designed for patients with MNM. The QoLNMD is short enough to be used in clinical practice (26 items).

The next step was to validate the QoLNMD reassessing its psychometric properties in a new patient sample and calibrate the IRR measurement system. The purpose of these new part of study was to validate the French version of the QoL-NMD on a confirmatory sample of patients and to calibrate its measurement system.

A prospective study in 8 NMD referral centers (France) was conducted. Both the QoL-NMD and a validated generic questionnaire (the WHOQOLBREF) were administered to patients. Confirmatory psychometric analyses were performed on the new sample while the Items Response Theory (IRT) model calibration was performed on all patients ever recruited using the Partial Credit Model (Rasch).

156 patients were included for the confirmatory psychometric analysis. All three domains showed adequate psychometric properties (internal consistency: repeatability ; scalability) and met IRT assumptions. The IRT model calibration was performed successfully on 315 patients. Minimum detectable change estimates are distribution based and should be verified by external meaningful anchors.

ELIGIBILITY:
Inclusion Criteria:

* Patient with neuromuscular disease

Exclusion Criteria:

* <18 yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French Patients, young adults and adults, with a diagnosed neuromuscular disease, of any known form.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2006-06; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Self reported form of items measuring the Quality of Life | 0 month
  The Quality of Life questionnaire used is QoLNMD

SECONDARY OUTCOMES:
Self reported form of items measuring the Quality of Life | 6 months
  The Quality of Life questionnaire used is QoLNMD
Self reported form of items measuring the Quality of Life | 1 year
  The Quality of Life questionnaire used is QoLNMD

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France